CLINICAL TRIAL: NCT01630629
Title: "Bone Density and Calcitropic Hormones During Lactation in African-American and Caucasian Women"
Brief Title: Longitudinal Lactation Bone Density Study
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Mara Horwitz, Associate Professor of Medicine, University of Pittsburgh
Other Study IDs: PRO12050600
Record Dates: First submitted 2012-06-20; First posted 2012-06-28 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Lactation; Other Disorders of Bone Density and Structure; Endocrine; Complications
Keywords: Lactation; Weaning; Bone Density; Endocrine; Physiological Properties; Bone Metabolism
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and breast milk
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- African-American Lactating Women: Healthy African-American women who are exclusively breast-feeding.
- Caucasian Lactating Women: Healthy Caucasian women who are exclusively breast-feeding.

SUMMARY:
Changes in maternal calcium metabolism are necessary during lactation to provide adequate calcium in breast milk for development of the newborn skeleton. The calcium in milk is derived from the maternal skeleton, resulting in significant bone loss, a process thought to be mediated by the actions of parathyroid hormone-related protein (PTHrP) in combination with a decreased estrogen levels. After weaning, bone lost during lactation is rapidly regained.

Differences between African-American and Caucasian bone metabolism are well documented and include higher bone mineral density (BMD), lower risk of fragility fracture, lower 25-hydroxyvitamin D (25(OH) D), and higher PTH in African-Americans compared to Caucasians. Most studies of bone metabolism in lactating women have been done in Caucasians. Because of differences in bone metabolism between African-Americans and Caucasians, we do not know whether African-Americans will have similar findings.

The primary aim of this study is to compare the changes in bone mineral density (BMD) during lactation in African-Americans with those in Caucasians. It is not known whether the loss in BMD during lactation will be the same for both races. African-Americans display skeletal resistance to PTH with short-term infusions and have lower bone resorption, higher BMD and lower fracture risk than Caucasians. A recent study by our group indicated that lactating African-American mothers had slightly lower bone resorption but quantitatively similar bone formation compared to Caucasians. However, there was a significant increase of 2-3 fold in markers of bone formation and resorption in both groups. Therefore, it is currently not known whether the loss in BMD during lactation will be the same for both races. Primary outcome measures in this study will include spine, hip and radius BMD by Dual X-Ray Absorbiometry (DXA)Scans during lactation (at 2,12 and 24 weeks postpartum or at weaning if prior to 24 weeks postpartum, and six months after weaning (+1 week). This longitudinal protocol will distinguish between two hypotheses. Either: a) as measured by BMD, bone loss in African-Americans during lactation will be equal to that in Caucasians, and skeletal recovery will be the same or possibly accelerated compared to Caucasians; or, b) African-Americans will be resistant to bone loss during lactation compared to Caucasians because of resistance to Parathyroid Hormone-related Protein (PTHrP).

DETAILED DESCRIPTION:
Pregnancy and lactation are both states of altered maternal calcium metabolism. Maternal calcium mobilization is essential in the provision of an adequate calcium supply to the developing fetus and infant. During pregnancy approximately 30 grams of calcium is required for fetal skeletal development. The extra calcium is derived mostly from increased maternal intestinal absorption, mediated by 1,25 dihydroxyvitamin D (1). During lactation, it is estimated that 600-1000 ml of milk are produced daily with a net maternal calcium loss of 200-400 mg per day (2,3). This calcium is derived from the maternal skeleton, resulting in bone loss of as much as 10% of trabecular bone with serial bone density measurements (3). Demineralization is thought to be mediated predominantly by the actions of parathyroid hormone-related protein (PTHrP) in combination with a suppressed estrogen state. Interestingly, this state rapidly reverses itself with weaning (4,5). Several studies have shown that initial PTHrP measurements are significantly higher in lactating women(3). PTHrP in lactation is produced in high amounts by the mammary gland. Once in the circulation, PTHrP increases bone resorption from the maternal skeleton and increases calcium resorption at the level of the kidney (5,6,27). PTHrP levels have been found to be elevated as much as 10,000 fold in milk as compared with maternal serum, and further increase with suckling (1,6,28). In mouse models, tissue specific-ablation of the PTHrP gene in lactating mammary gland results in decreased bone loss(6).

Given the rapid bone loss reported in lactation, an increase in markers of bone resorption and a decrease in markers of bone formation might be expected. However, a recently published study by our group showed that both markers of bone formation and bone resorption were significantly elevated in lactating Caucasian women (7). This seems unlikely as tight coupling of bone formation and resorption would not result in net calcium mobilization and rapid bone loss during lactation. A more likely explanation is that while bone resorption markers accurately reflect robust osteoclastic bone resorption, the increase in markers of bone formation reflects an increase in immature, partially differentiated pre-osteoblasts that are arrested in development and therefore unable to effectively form new bone. Thus, the rate of resorption exceeds that of formation during lactation and results in a temporary net loss. To support this idea, rat studies have shown that continuous exposure to PTH and PTHrP recruits and initiates osteoblast differentiation, but stops the program prematurely at the preosteoblast transition (8,9,10). This would also suggest a mechanism for the rapid recovery seen after weaning: after withdrawing the PTHrP stimulus, osteoclast-mediated bone resorption would abruptly cease, and previously recruited osteoblast precursors would rapidly complete their differentiation program and restore bone lost during lactation.

African-American bone metabolism differs from Caucasian bone metabolism in several ways. African-Americans display higher bone density and are at lower risk of developing osteoporosis and osteoporotic fracture compared to Caucasians (15-17,29-31). There are may factors which may explain these racial differences in bone metabolism, including altered calcium economy, vitamin D differences, peak attained bone mass, muscle mass and obesity, remodeling rates, bone micro-architecture, hip axis geometry , and other unknown hereditary differences. In particular, it is well established that 25-Hydroxyvitamin D (25-OH D) levels are much lower in African-Americans, due to darker pigmentation resulting in reduced dermal production of 25-OH D as well as reduced intake of vitamin D (11). This hypovitaminosis results in a relative secondary hyperparathyroidism, corroborated by higher levels of PTH and 1,25 dihydroxyvitamin D as well as decreased urinary calcium excretion (12-14). Paradoxically, these higher PTH levels do not correlate with an increase in bone loss. In fact, bone turnover is actually reduced compared to Caucasians, suggesting that African-American bones are more resistant to the effects of PTH, whereas renal sensitivity is maintained or increased (14,18).

The vast majority of studies examining bone metabolism in lactating women have been in Caucasian women. Studies on bone turnover and calcitropic hormones in lactating African-Americans are scarce. Over ten years ago, a study examined markers of bone metabolism in a population of lactating Gambian women (in Gambia) and compared them with a similar cohort of British lactating women (in the UK). The study demonstrated significant increases in older markers of bone formation and resorption during lactation, but also showed higher levels of PTH, 1,25 Vitamin D, serum phosphate, osteocalcin, and alkaline phosphatase in the Gambian lactating population compared with the British lactating population (19). However, Gambian women differ significantly from black women in the developed world in terms of nutrition, both overall calories and calcium intake. Also in contrast to African-Americans, black Gambian women displayed lower BMD than Caucasians. Interestingly, in these studies, Gambian women demonstrated significant losses in whole body and hip BMD during lactation and showed little evidence of bone mass regain after weaning. In fact, Gambian women had continued BMD loss at the hip, in contrast to Caucasian controls.

A recent study by our group (unpublished) explored bone turnover markers and calcium metabolism in African-American lactation. Markers of bone resorption were lower in African-American than Caucasians in non-lactating young women, but increased 2-3 fold in both groups during lactation. Baseline bone formation was comparable in African-Americans and Caucasians, also increasing 2-3 fold in both groups. Fractional excretion of calcium was lower in African-Americans at baseline and remained constant in both groups during lactation. It remains unclear whether bone loss occurs at a similar rate during lactation in the African-American population.

Up to this point, there have been no studies in African-Americans that have utilized bone densitometry to quantitate bone loss and recovery during lactation. This study aims to demonstrate changes in bone density in African-American women during the high bone turnover state of lactation. It will also permit measurements of calcium metabolism, markers of bone formation and resorption, and calcitropic hormones to be compared to bone density changes. We will also look for racial differences in lactating bone metabolism by directly comparing a cohort of African-American lactating women with a similar Caucasian cohort. No prior studies have been done comparing bone mineral density changes in lactating American black and Caucasian women.

ELIGIBILITY:
Inclusion Criteria:

* 21-45 years old
* Post-partum after a singleton pregnancy
* Exclusively breast-feeding (not more than one supplemental bottle of formula per day)
* African-American or Caucasian by self-identification

Exclusion Criteria:

* Subjects with cardiac, hypertensive, vascular, renal (serum creatinine of >1.5), pulmonary, endocrine, musculoskeletal, hepatic, hematologic, malignant or rheumatologic disease
* Fractures or bone surgery within the past 12 months
* Smokers and subjects with history of significant alcohol or drug use
* Pregnant women
* Women who achieved pregnancies with IVF or other hormonal manipulation
* Women who had significant complications with the most recent pregnancy or who are unable to exclusively breastfeed beginning at birth
* Subjects on chronic medications other than
* stable doses of thyroid hormone
* oral contraceptives
* vitamin supplements
* Women on Depo-Provera will be excluded
* Receiving an investigational drug within 90 days
* Weight greater than 130 kg
* Z-score -3.0 or less (hip or spine) on initial DXA

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: New mothers will be recruited from UPMC hospital population, primarily Magee Womens Hospital. As this is a study which aims to describe racial differences in bone metabolism during lactation in African-Americans and Caucasians, subjects must identify themselves as belonging to one of these groups.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2012-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in bone density measurements (BMD) | Change from baseline in BMD at 2,12, 24 weeks postpartum, and six months after weaning.
  Primary outcome measures will include spine, hip and radius BMD by DXA at 2, 12, and 24 weeks post-partum and 6 months post-weaning.

SECONDARY OUTCOMES:
Change from baseline of bone metabolism measurements | Change from baseline at 2, 12,and 24 weeks postpartum, and six months after weaning.
  Bone metabolism measurements include: markers of bone turnover including calcium metabolic parameters such as calcium, phosphorus, fractional excretion of calcium, PTH(1-84), PTHrP, vitamin D metabolites, estradiol, sex hormone binding globulin (SHBG), prolactin, and breast milk calcium levels.

CONTACTS AND LOCATIONS:
Overall Officials: Mara Horwitz, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kovacs CS. Calcium and bone metabolism during pregnancy and lactation. J Mammary Gland Biol Neoplasia. 2005 Apr;10(2):105-18. doi: 10.1007/s10911-005-5394-0. PMID 16025218
- [Background] Sowers MF, Hollis BW, Shapiro B, Randolph J, Janney CA, Zhang D, Schork A, Crutchfield M, Stanczyk F, Russell-Aulet M. Elevated parathyroid hormone-related peptide associated with lactation and bone density loss. JAMA. 1996 Aug 21;276(7):549-54. PMID 8709404
- [Background] Kovacs CS, Kronenberg HM. Maternal-fetal calcium and bone metabolism during pregnancy, puerperium, and lactation. Endocr Rev. 1997 Dec;18(6):832-72. doi: 10.1210/edrv.18.6.0319. No abstract available. PMID 9408745
- [Background] Sowers M, Eyre D, Hollis BW, Randolph JF, Shapiro B, Jannausch ML, Crutchfield M. Biochemical markers of bone turnover in lactating and nonlactating postpartum women. J Clin Endocrinol Metab. 1995 Jul;80(7):2210-6. doi: 10.1210/jcem.80.7.7608281.
- [Background] VanHouten JN, Wysolmerski JJ. Low estrogen and high parathyroid hormone-related peptide levels contribute to accelerated bone resorption and bone loss in lactating mice. Endocrinology. 2003 Dec;144(12):5521-9. doi: 10.1210/en.2003-0892. Epub 2003 Sep 18. PMID 14500568
- [Background] VanHouten JN, Dann P, Stewart AF, Watson CJ, Pollak M, Karaplis AC, Wysolmerski JJ. Mammary-specific deletion of parathyroid hormone-related protein preserves bone mass during lactation. J Clin Invest. 2003 Nov;112(9):1429-36. doi: 10.1172/JCI19504. PMID 14597768
- [Background] Carneiro RM, Prebehalla L, Tedesco MB, Sereika SM, Hugo M, Hollis BW, Gundberg CM, Stewart AF, Horwitz MJ. Lactation and bone turnover: a conundrum of marked bone loss in the setting of coupled bone turnover. J Clin Endocrinol Metab. 2010 Apr;95(4):1767-76. doi: 10.1210/jc.2009-1518. Epub 2010 Feb 11. PMID 20150580
- [Background] Wang YH, Liu Y, Buhl K, Rowe DW. Comparison of the action of transient and continuous PTH on primary osteoblast cultures expressing differentiation stage-specific GFP. J Bone Miner Res. 2005 Jan;20(1):5-14. doi: 10.1359/JBMR.041016. Epub 2004 Oct 25. PMID 15619664
- [Background] Dobnig H, Turner RT. The effects of programmed administration of human parathyroid hormone fragment (1-34) on bone histomorphometry and serum chemistry in rats. Endocrinology. 1997 Nov;138(11):4607-12. doi: 10.1210/endo.138.11.5505. PMID 9348185
- [Background] van der Horst G, Farih-Sips H, Lowik CW, Karperien M. Multiple mechanisms are involved in inhibition of osteoblast differentiation by PTHrP and PTH in KS483 Cells. J Bone Miner Res. 2005 Dec;20(12):2233-44. doi: 10.1359/JBMR.050821. Epub 2005 Aug 29. PMID 16294276
- [Background] Cosman F, Nieves J, Dempster D, Lindsay R. Vitamin D economy in blacks. J Bone Miner Res. 2007 Dec;22 Suppl 2:V34-8. doi: 10.1359/jbmr.07s220. PMID 18290719
- [Background] Harris SS, Soteriades E, Dawson-Hughes B; Framingham Heart Study; Boston Low-Income Elderly Osteoporosis Study. Secondary hyperparathyroidism and bone turnover in elderly blacks and whites. J Clin Endocrinol Metab. 2001 Aug;86(8):3801-4. doi: 10.1210/jcem.86.8.7783. PMID 11502814
- [Background] Bell NH, Yergey AL, Vieira NE, Oexmann MJ, Shary JR. Demonstration of a difference in urinary calcium, not calcium absorption, in black and white adolescents. J Bone Miner Res. 1993 Sep;8(9):1111-5. doi: 10.1002/jbmr.5650080912. PMID 8237481
- [Background] Fuleihan GE, Gundberg CM, Gleason R, Brown EM, Stromski ME, Grant FD, Conlin PR. Racial differences in parathyroid hormone dynamics. J Clin Endocrinol Metab. 1994 Dec;79(6):1642-7. doi: 10.1210/jcem.79.6.7989469.
- [Background] Nelson DA, Jacobsen G, Barondess DA, Parfitt AM. Ethnic differences in regional bone density, hip axis length, and lifestyle variables among healthy black and white men. J Bone Miner Res. 1995 May;10(5):782-7. doi: 10.1002/jbmr.5650100515. PMID 7639113
- [Background] George A, Tracy JK, Meyer WA, Flores RH, Wilson PD, Hochberg MC. Racial differences in bone mineral density in older men. J Bone Miner Res. 2003 Dec;18(12):2238-44. doi: 10.1359/jbmr.2003.18.12.2238. PMID 14672360
- [Background] Thomas PA. Racial and ethnic differences in osteoporosis. J Am Acad Orthop Surg. 2007;15 Suppl 1:S26-30. doi: 10.5435/00124635-200700001-00008. PMID 17766786
- [Background] Cosman F, Morgan DC, Nieves JW, Shen V, Luckey MM, Dempster DW, Lindsay R, Parisien M. Resistance to bone resorbing effects of PTH in black women. J Bone Miner Res. 1997 Jun;12(6):958-66. doi: 10.1359/jbmr.1997.12.6.958. PMID 9169356
- [Background] Prentice A, Jarjou LM, Stirling DM, Buffenstein R, Fairweather-Tait S. Biochemical markers of calcium and bone metabolism during 18 months of lactation in Gambian women accustomed to a low calcium intake and in those consuming a calcium supplement. J Clin Endocrinol Metab. 1998 Apr;83(4):1059-66. doi: 10.1210/jcem.83.4.4737. PMID 9543117
- [Background] Horwitz MJ, Tedesco MB, Sereika SM, Hollis BW, Garcia-Ocana A, Stewart AF. Direct comparison of sustained infusion of human parathyroid hormone-related protein-(1-36) [hPTHrP-(1-36)] versus hPTH-(1-34) on serum calcium, plasma 1,25-dihydroxyvitamin D concentrations, and fractional calcium excretion in healthy human volunteers. J Clin Endocrinol Metab. 2003 Apr;88(4):1603-9. doi: 10.1210/jc.2002-020773. PMID 12679445
- [Background] Stewart AF, Vignery A, Silverglate A, Ravin ND, LiVolsi V, Broadus AE, Baron R. Quantitative bone histomorphometry in humoral hypercalcemia of malignancy: uncoupling of bone cell activity. J Clin Endocrinol Metab. 1982 Aug;55(2):219-27. doi: 10.1210/jcem-55-2-219. PMID 7085851
- [Background] Finkelstein JS, Lee ML, Sowers M, Ettinger B, Neer RM, Kelsey JL, Cauley JA, Huang MH, Greendale GA. Ethnic variation in bone density in premenopausal and early perimenopausal women: effects of anthropometric and lifestyle factors. J Clin Endocrinol Metab. 2002 Jul;87(7):3057-67. doi: 10.1210/jcem.87.7.8654. PMID 12107201
- [Background] Perry HM 3rd, Horowitz M, Morley JE, Fleming S, Jensen J, Caccione P, Miller DK, Kaiser FE, Sundarum M. Aging and bone metabolism in African American and Caucasian women. J Clin Endocrinol Metab. 1996 Mar;81(3):1108-17. doi: 10.1210/jcem.81.3.8772584.
- [Background] Horwitz MJ, Tedesco MB, Sereika SM, Syed MA, Garcia-Ocana A, Bisello A, Hollis BW, Rosen CJ, Wysolmerski JJ, Dann P, Gundberg C, Stewart AF. Continuous PTH and PTHrP infusion causes suppression of bone formation and discordant effects on 1,25(OH)2 vitamin D. J Bone Miner Res. 2005 Oct;20(10):1792-803. doi: 10.1359/JBMR.050602. Epub 2005 Jun 6. PMID 16160737
- [Background] Kalkwarf HJ, Specker BL, Ho M. Effects of calcium supplementation on calcium homeostasis and bone turnover in lactating women. J Clin Endocrinol Metab. 1999 Feb;84(2):464-70. doi: 10.1210/jcem.84.2.5451. PMID 10022402
- [Background] Nelson DA, Barondess DA, Hendrix SL, Beck TJ. Cross-sectional geometry, bone strength, and bone mass in the proximal femur in black and white postmenopausal women. J Bone Miner Res. 2000 Oct;15(10):1992-7. doi: 10.1359/jbmr.2000.15.10.1992. PMID 11028452
- [Background] Syed MA, Horwitz MJ, Tedesco MB, Garcia-Ocana A, Wisniewski SR, Stewart AF. Parathyroid hormone-related protein-(1--36) stimulates renal tubular calcium reabsorption in normal human volunteers: implications for the pathogenesis of humoral hypercalcemia of malignancy. J Clin Endocrinol Metab. 2001 Apr;86(4):1525-31. doi: 10.1210/jcem.86.4.7406. PMID 11297578
- [Background] Burtis WJ, Brady TG, Orloff JJ, Ersbak JB, Warrell RP Jr, Olson BR, Wu TL, Mitnick ME, Broadus AE, Stewart AF. Immunochemical characterization of circulating parathyroid hormone-related protein in patients with humoral hypercalcemia of cancer. N Engl J Med. 1990 Apr 19;322(16):1106-12. doi: 10.1056/NEJM199004193221603. PMID 2320080
- [Background] Luckey MM, Wallenstein S, Lapinski R, Meier DE. A prospective study of bone loss in African-American and white women--a clinical research center study. J Clin Endocrinol Metab. 1996 Aug;81(8):2948-56. doi: 10.1210/jcem.81.8.8768857.
- [Background] Cauley JA, Wampler NS, Barnhart JM, Wu L, Allison M, Chen Z, Hendrix S, Robbins J, Jackson RD; Women's Health Initiative Observational Study. Incidence of fractures compared to cardiovascular disease and breast cancer: the Women's Health Initiative Observational Study. Osteoporos Int. 2008 Dec;19(12):1717-23. doi: 10.1007/s00198-008-0634-y. Epub 2008 Jul 16. PMID 18629572
- [Background] Cauley JA, Palermo L, Vogt M, Ensrud KE, Ewing S, Hochberg M, Nevitt MC, Black DM. Prevalent vertebral fractures in black women and white women. J Bone Miner Res. 2008 Sep;23(9):1458-67. doi: 10.1359/jbmr.080411. PMID 18442309